CLINICAL TRIAL: NCT00455871
Title: An Open-Label, Single-Site, Comparative, Pilot Study of the Treatment Effects of Combination Therapy of Lucentis (Ranibizumab) Plus Reduced Fluence Photodynamic Therapy With Visudyne in Patients With Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Study of Treatment Effects of Combination Therapy of Lucentis Plus Reduced Fluence PDT With Visudyne in Patients With Exudative AMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barnes Retina Institute (Other)
Collaborators: QLT Inc. (Industry)
Responsible Party: Gaurav Shah, M.d., Barnes Retina Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0769; NCT00455871
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Age-Related Macular Degeneration
Keywords: macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Verteporfin; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lucentis plus Reduced Fluence PDT same day (Active Comparator)
  Interventions: Drug: reduced fluence photodynamic therapy with Visudyne; Drug: Lucentis
- Lucentis plus reduced fluence PDT 1-2 weeks later (Active Comparator)
  Interventions: Drug: reduced fluence photodynamic therapy with Visudyne; Drug: Lucentis

INTERVENTIONS:
Drug: reduced fluence photodynamic therapy with Visudyne — reduced fluence photodynamic therapy with visudyne
Drug: Lucentis — Lucentis intravitreal injection

SUMMARY:
The purpose of this study is to determine the benefits, if any, of combination therapy with Lucentis plus reduced fluence photodynamic therapy with Visudyne.

DETAILED DESCRIPTION:
The study will have two treatment groups. Each group will receive intravitreal injections (injection of medication in the jelly-like part of the back of the eye). One group (Group1) of approximately 15 patients will receive 0.5 mg of Lucentis™ followed by reduced fluence Photodynamic Therapy (PDT) with Visudyne ® 1-2 weeks later. The other group (Group 2) of approximately 15 patients will receive 0.5 mg of Lucentis™ followed by Photodynamic Therapy with Visudyne on the same day. patients will be assigned at random to receive one of the two treatments arms in the study. The dose received at the first injection will be the same dose received throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Treatment- naïve patients with active, subfoveal, exudative AMD
* Patients with visual acuity of 20/40-20/320 in the study eye
* Subfoveal choroidal neovascularization (CNV) must be at least 50% of the total lesion size Total area of lesion components other that CNV must be less than 50% of the total lesion size
* The lesion must be < 5400microns in greatest linear dimension (GLD)
* Lesion size < 10 DA
* Occult with no classic CNV lesions must have presumed recent disease progression:

  1. Blood associated with the lesion at baseline
  2. Loss of visual acuity in the previous 3 months: a: > 5 letter loss (ETDRS equivalent) or b: 2 or more lines using a snellen or equivalent chart
  3. > 10% increase in GLD as assessed by fluorescein angiography in the previous 3 months
* Previous treatment for CNV with anti-VEGF agents, intraocular steroids and/or Photodynamic therapy with Visudyne® in the study eye
* Geographic atrophy or fibrosis in the study eye
* Intraocular surgery within 6 weeks of enrollment
* Subretinal hemorrhage > 50% of the total lesion
* Patients with intraocular pressure greater than 30 mm/Hg on 2 pressure-lowering medications
* Patients with severe disciform scarring.
* Inability to make study visits
* Advanced glaucoma
* Allergies to porfins or a known hypersensitivity to any component of Visudyne®
* Patients with porphyria
* Pregnancy or lactation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of the combination therapy | 12 months and 24 months
To assess efficacy of the two timing regimens | 12 months and 24 months

SECONDARY OUTCOMES:
To evaluate the number of Lucentis injections and the number of PDT treatments required during the study | 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav K. Shah, MD, Principal Investigator — Barnes Retina Institute
Locations (1):
- Barnes Retina Institute, St Louis, Missouri, United States